CLINICAL TRIAL: NCT02637843
Title: Randomized Comparison of Coated Slender Versus Un-coated Traditional Sheath
Brief Title: Randomized Comparison of Sheaths for Radial Access
Acronym: ACCESS-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, MD, DmSc, Associate professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ACCESS-I
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Radial Angiography
Keywords: radial; angiography; angioplasty; randomized; sheath; slender

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slender arm (Active Comparator): Uses the terumo slender sheath for radial angiography or angioplasty
  Interventions: Device: Slender Sheath
- Standard arm (No Intervention): Uses the terumo standard sheath (Routine) for radial angiography or angioplasty

INTERVENTIONS:
Device: Slender Sheath — Comparing outcomes for two different sheaths used during radial CAG/PCI
  Arms: Slender arm

SUMMARY:
Coronary angiography (CAG) and possible angioplasty (Percutaneous Coronary Intervention = PCI) can be performed by access from the groin (a. femoralis), the wrist (a. radialis) or the elbow (a. brachialis). It is well established that there is less risk of bleeding complications when using a radial access. The smaller diameters of the vessels in the forearm, however, may result in increased risk of pain during CAG/PCI via a. radialis. This is associated with vascular spasm (spasm tendency). Ultimately this means that one may have to convert to access via a. femoralis.

To perform a CAG/PCI, a tube (a so-called sheath) has to be inserted in a. radialis. It is unclear whether the design of the sheaths can reduce the spasm tendency, thus reducing pain. Terumo has recently introduced a new kind of sheath, so-called Terumo Glide Slender Heath Coated (hereafter referred to as "Slender sheath"). This sheath is partly coated, partly made of a thinner material. "Slender sheath" thus has an outer diameter smaller than that of the sheath from traditional use (Terumo Radio Focus sheath, hereafter referred to as "Standard sheath"), although the inner diameter (lumen) is the same in the two sheaths. In turn, the "Slender sheath" is more fragile and far more expensive.

The purpose of the present study is to evaluate whether use of slender sheath compared with standard sheath is Associated with less pain and fewer complications following CAG/PCI.

DETAILED DESCRIPTION:
Study design: Randomized study

Purposes: to investigate whether the use of "Slender sheath" is associated with less pain compared to use of "Standard Sheath" and less complications corresponding at the access site. Specific hypotheses:

1. Use of "Slender sheath" results in less pain related to CAG/PCI compared to use of "Standard sheath".
2. Use of "Slender sheath" is associated with fewer conversions to femoral access compared to use of "Standard sheath".
3. Use of "Slender sheath" is associated with less use of analgesic during the procedure compared to use of "Standard sheath".
4. Use of "Slender sheath" is associated with fewer cases of occlusion of a. radialis at discharge and post-examination compared to use of "Standard sheath".

Time Schedule The trial will run from December 2015 until a total number of 1000 patients are included. It is expected that the data collection and publication of the results will be completed within a year.

Endpoints

1. Pain related to the application of the sheath (Visual Analog Scale = VAS)
2. Maximal pain during CAG/PCI (VAS)
3. Frequency of conversions to femoral access
4. Use of analgesics (cumulative amount of mg Fentanyl given)
5. Use of sedatives (cumulative amount of mg Midazolam given)
6. Use of Verapamil (cumulative amount of mg given, used to reduce spasms)
7. Number of catheters used
8. Number of sheaths used (femoral and radial)
9. Occlusion of a. radialis at the time of discharge estimated by ultrasound of the artery
10. Occlusion of a. radialis after a month (Assumes that all patients with open vessels at discharge also have open vessels after a month. Only patients with occluded vessels at discharge will be offered a new ultrasound scan)

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for radial angiography or angioplasty
* Able to give written informed consent

Exclusion Criteria:

* Negative Barbaue test or Allens test
* Use of 8F catheters

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pain during sheath insertion | 1-2 minutes during sheath insertion
  Maximal pain (Visual analogue scale) during sheath insertion
Pain during the procedure | 10 minutes to 2 hours (during CAG/PCI)
  Maximal pain (Visual analogue scale) during CAG/PCI
Proportion converted to femoral access | 10 minutes to 2 hours (during CAG/PCI)
  Proportion of patients where the operator has to change to femoral access to complete the CAG/PCI
Use of analgesics, sedatives and verapamil during the procedure | 10 minutes to 2 hours (during CAG/PCI)
  cumulative amount of analgesics, sedatives and verapamil during the procedure
Patency of a.radialis | Within one month of CAG/PCI
  Ultrasound and reverse Barbaeu test is performed to test patency of a.radialis following CAG/PCI. If patency not documented at time of discharge the tests are repeated at one month. The artery is patent if normal Barbaue test and ultrasound without occlusion.

SECONDARY OUTCOMES:
Number of catheters used | 10 minutes to 2 hours (during CAG/PCI)
  cumulative number of catheters used during the procedure
Number of sheaths used | 10 minutes to 2 hours (during CAG/PCI)
  cumulative number of sheaths used during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Aarhus University Hospital in Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No